CLINICAL TRIAL: NCT00356915
Title: A Phase III Randomized, Evaluator-Blind, Parallel Group Study of the Safety and Efficacy of Itraconazole Tablets, Itraconazole Capsules and Placebo in the Treatment of Onychomycosis of the Toenail.
Brief Title: Itraconazole Tablets Vs. Itraconazole Capsules vs. Placebo in Onychomycosis of the Toenail.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT0300-302-INT
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2012-01-04 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Onychomycosis
Keywords: Nail fungus; Onychomycosis; Itraconazole; Toenail
MeSH Terms: conditions — Onychomycosis | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Itraconazole tablets (Experimental): Itraconazole 200 mg tablets
  Interventions: Drug: Itraconazole 200mg tablets
- Itraconazole capsules (Active Comparator): Two Itraconazole 100 mg capsules were taken daily.
  Interventions: Drug: Itraconazole 100mg capsules
- Placebo tablets (Placebo Comparator): The itraconazole 200-mg tablets and placebo tablets exactly matched one another and were white to slightly grey in color, were oblong and biconvex in shape, and were melt-extrusion, film-coated.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Itraconazole 100mg capsules — Subjects took two 100mg capsules once per day after a full meal. The dose dose was taken the day before the Week 12 visit.
  Other Names: Sporanox®
  Arms: Itraconazole capsules
Drug: Itraconazole 200mg tablets — Subjects took one 200mg tablet once per day after a full meal. The last dose was taken the day before the Week 12 visit.
  Other Names: Onmel
  Arms: Itraconazole tablets
Drug: Placebo tablets — Placebo tablets are the same as the Itraconazole tablets but without the active drug included. Subjects took one tablet once per day after a full meal. The last tablet was taken the day before the Week 12 visit.
  Other Names: placebo
  Arms: Placebo tablets

SUMMARY:
Onychomycosis is a common condition accounting for approximately half of all nail disorders. It is most commonly caused by dermatophytes. Itraconazole has been approved for the treatment of onychomycosis in the United States with an approved dosage regimen for the treatment of onychomycosis of the toenail of once daily (QD) treatment with 200mg of itraconazole (two 100 mg capsules) for 12 weeks. Barrier Therapeutics has developed a 200 mg tablet which could be used in a more convenient one-tablet-per-day dosing regimen. This clinical trial will compare the efficacy and safety of this new tablet formulation with itraconazole capsules and placebo.

DETAILED DESCRIPTION:
Onychomycosis is common and accounts for about half of all nail disorders. Usually the cause is due to dermatophytes, either Trichophyton rubrum (71%) or Trichophyton mentagrophytes (20%) but may also be due to yeast infection, usually Candida albicans.

The prevalence of onychomycosis in the United States population as a whole is 13% and is more prevalent in the elderly (60%). Onychomycosis of the toenail recurs and is thought to have a genetic component.

Onychomycosis can result in permanent nail deformity. This disease has a significant impact on the patient's quality of life (e.g., concern with the appearance of the toenails and fingernails, interference with wearing shoes, walking and sports activities).

Itraconazole has been approved for the treatment of onychomycosis in the United States since the mid-nineteen-nineties. The approved dosage regimen for treatment of onychomycosis of the toenail is once daily (QD) treatment with 200 mg of itraconazole (Sporanox®, Janssen Pharmaceutical Products, L.P., Titusville, NJ, USA) for 12 weeks. The approved dosage form is a 100mg capsule. Barrier Therapeutics has developed a 200mg tablet which could be used in a more convenient one-tablet-per-day dosing regimen.

This clinical trial will compare the efficacy and safety of this new tablet formulation with itraconazole capsules and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of onychomycosis of at least one great toenail
* Percent Nail Involvement Score of the more severely affected great toenail (the Target Toenail) must be between 2 and 3 (25-75% of the nail unit).
* Length of Unaffected Part of the Target Toenail ≥2mm
* Direct microscopic examination with KOH that is positive for the hyphae associated with dermatophytes on the target toenail
* Subjects must have signed informed consent
* If the subject is woman of childbearing potential, she must have a negative urine pregnancy test and agree to use an effective form of birth control until the first menses after 60 days following the last dose of study medication.

Exclusion Criteria:

* Onychomycosis caused by Candida spp. without the presence of a dermatophyte
* Participation in a clinical trial for the systemic treatment of onychomycosis of the toenail within 24 weeks prior to Visit 1
* Use of systemic antifungals within 12 weeks prior to Visit 1
* Use of topical antifungal nail lacquer within 30 days prior to Visit 1
* Use of any other topical onychomycosis treatment on any toenail within 7 days prior to Visit 1
* Evidence of ventricular dysfunction such as congestive heart failure (CHF) or a history of CHF
* Known liver disease or a history of liver toxicity with other drugs
* Use of systemic immunosuppressants

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1381 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (68):
- United States (52):
  - Radiant Research -Birmingham, Birmingham, Alabama
  - University of Alabama School of Medicine, Birmingham, Alabama
  - Radiant Research - Tucson, Tuscon, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - East Bay Dermatology Medical Group Inc., Fremont, California
  - Skin Surgey Medical Group, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - University of California, San Francisco, California
  - Radiant Research - Santa Rosa, Santa Rosa, California
  - Meridian Skincare, Englewood, Colorado
  - The Savin Center, New Haven, Connecticut
  - Dr. Stephen Horwitz, Aventure, Florida
  - International Dermatology Research Inc., Miami, Florida
  - FMX Research Corporation, Miami, Florida
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Radiant Research - St. Petersburg, St. Petersburg, Florida
  - Radiant Research - West Palm Beach, West Palm Beach, Florida
  - Radiant Research - Atlanta West, Austell, Georgia
  - Gwinnett Clinical Research Center Inc., Snellville, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Radiant Research - Chicago, Chicago, Illinois
  - Radiant Research - Kansas City, Overland Park, Kansas
  - Dr. David Fivenson, Ann Arbour, Michigan
  - Skin and Vein Center, Troy, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - VA Medical Center, Minneapolis, Minnesota
  - Dr. Eduardo Tschen, Albuquerque, New Mexico
  - Skin Specialty Group, New York, New York
  - Columbia University Medical Center, New York, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Dermatology Clinical Research Center, Cincinnati, Ohio
  - Radiant Research - Cincinnati, Cincinnati, Ohio
  - Northwest Cutaneous Research, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiant Research - Anderson, Anderson, South Carolina
  - Radiant Research - Greenville, Greenville, South Carolina
  - Dr. J. M. Humeniuk, Greer, South Carolina
  - Dermatology East, Germantown, Tennessee
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch Inc., Austin, Texas
  - Dr. Terry Jones, Bryan, Texas
  - Radiant Research - Dallas North, Dallas, Texas
  - Dr. Stephen Miller, San Antoinio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - South Valley Dermatology Center, West Jordan, Utah
  - Pariser Dermatology Specialists Ltd., Norfolk, Virginia
  - Radiant Research - Tacoma, Tacoma, Washington
  - Madison Skin and Research Inc., Madison, Wisconsin
  - Advanced Healthcare S. C., Milwaukee, Wisconsin
- Canada (8):
  - Dr. Kirk Barber, Calgary, Alberta
  - Dr. Richard Thomas, Vancouver, British Columbia
  - Dr. Marc Bourcier, Moncton, New Brunswick
  - Dr. Aditja Gupta, London, Ontario
  - Dr. Chuck Lynde, Markham, Ontario
  - EntraLogix, Oakville, Ontario
  - Dr. Jerry Tan, Windsor, Ontario
  - Dr. Robert Bissonnette, Montreal, Quebec
- Edifico Professional Guarionex Lopez, Santo Domingo, Dominican Republic
- Dr. Manuel Briones, Guayaquil, Ecuador
- Centro Orquidea Blanca, San Pedro, Sula, Honduras
- Clinica Metropolis II, Panama City, Panama
- South Africa (4):
  - Langeberg Medical Centre, Cape Town
  - University of Cape Town, Cape Town
  - Dr. Z. F. Ahmed Vawda, Durban
  - DJW Navorsing, Krugerson

REFERENCES:
- [Derived] Maddin S, Quiring J, Bulger L. Randomized, placebo-controlled, phase 3 study of itraconazole for the treatment of onychomycosis. J Drugs Dermatol. 2013 Jul 1;12(7):758-63. PMID 23884486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from clinics in the US, Canada, South America, Ecuador, Dominican Republic, Panama, and Honduras.
Pre-assignment Details: Subjects were screened prior to randomization and had to have a positive result from a mycological culture of their toe nail (ie, culture that was positive for dermatophytes). If the culture was negative, they were not randomized to receive treatment and were discontinued from the study.
Groups:
- Itraconazole Tablets: Itraconazole 200 mg tablets. Subjects took one 200 mg tablet once per day after a full meal. The last dose was taken the day before the Week 12 visit.
- Itraconazole Capsules: Itraconazole 100 mg capsules
- Placebo Tablets: Tablets that were the same as the Itraconazole tables except that they did not contain the active drug (Itraconazole).
Period: Overall Study
Arm/Group | Itraconazole Tablets | Itraconazole Capsules | Placebo Tablets
Started | 593 | 590 | 198
Completed | 517 | 496 | 156
Not Completed | 76 | 94 | 42
Not completed — Non compliance | 1 | 2 | 1
Not completed — Protocol Violation | 2 | 3 | 2
Not completed — Withdrawal by Subject | 14 | 14 | 10
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 27 | 34 | 14
Not completed — Administrative Decision | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Adverse Event | 21 | 31 | 8
Not completed — Miscellaneous reasons | 11 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itraconazole Tablets | Itraconazole Capsules | Placebo Tablets | Total
Number analyzed (Participants) | 593 | 590 | 198 | 1381
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.86) | 47 (12.67) | 49.2 (11.12) | 47.4 (12.13)
Gender [Count of Participants; unit: Participants]
  Female | 441 | 440 | 153 | 1034
  Male | 152 | 150 | 45 | 347
Race/Ethnicity, Customized [Number; unit: Participants] — Subjects were permitted to select all choices from the list that apply to them with regard to race; ie, multiracial subjects would have checked more than one box and it would have been reported as such. Therefore the total number of subjects reported for race is greater than the number enrolled.
  Participants
    American Indian or Alaska Native | 7 | 7 | 4 | 18
    Asian | 5 | 4 | 2 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 48 | 48 | 18 | 114
    White | 512 | 493 | 169 | 1174
    Unknown or Not Reported | 25 | 41 | 7 | 73
Region of Enrollment [Number; unit: participants] — Participants were permitted to select all choices from the list that apply to them with regard to race; ie, multiracial participants would have checked more than one box and it would have been reported as such. Therefore the total number of participants reported for race is greater than the number enrolled.
  participants
    Panama | 9 | 9 | 3 | 21
    United States | 527 | 523 | 176 | 1226
    Canada | 23 | 21 | 8 | 52
    Ecuador | 6 | 8 | 3 | 17
    Honduras | 9 | 9 | 3 | 21
    Dominican Republic | 7 | 9 | 2 | 18
    South Africa | 12 | 11 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Mycological Cure of Target Toenail
Description: This study was designed to evaluate the superiority of itraconazole tablets to placebo tablets.
  Clinical Cure was defined as an IGA score of 0 for the target toenail; Mycological Cure was defined as a negative potassium hydroxide (KOH) exam and a negative culture for dermatophytes of the target toenail.
Time Frame: 1 year
Population: Intent to treat (ITT).
Measure: Number; unit: Percentage of participants
Groups:
- Itraconazole Tablets: Itraconazole 200mg tablets
Arm/Group | Itraconazole Tablets | Placebo Tablets
Number analyzed (Participants) | 593 | 198
Percentage of participants | 22.3 | 1
Statistical Analysis 1: Comparison: Itraconazole Tablets vs Placebo Tablets; P-Value from a Cochran-Mantel-Haenszel test, . The superiority analysis was restricted to the itraconazole 200-mg tablets and placebo tablets dosing groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; This was stratified by analysis center

2. Primary Outcome: Complete Cure - Itraconazole Tablets Compared to Itraconazole Capsules
Description: The primary efficacy endpoint was Compete Cure (consisting of a Clinical Cure and a Mycological Cure) at week 52. In this study, Clinical Cure was defined as an Investigator's Global Assessment (IGA) score of 0 for the target toenail; Mycological Cure was defined as a negative potassium hydroxide (KOH) examination and a negative culture outcome for dermatophytes of the target toenail. The efficacy analyses were conducted to demonstrate the non-inferiority of 1 itraconazole 200-mg tablet to 2 itraconazole 100-mg capsule.
Time Frame: 12 months
Population: Intent to treat (ITT).
Measure: Number; unit: Percentage of participants
Arm/Group | Itraconazole Tablets | Itraconazole Capsules | Placebo Tablets
Number analyzed (Participants) | 593 | 590 | 198
Percentage of participants | 22.3 | 21.7 | 1.0
Statistical Analysis 1: Comparison: Itraconazole Tablets vs Itraconazole Capsules; Comparison between the 2 itraconazole groups was based on lower bound of the 97.5% confidence interval for the difference. The non-inferiority analysis was restricted to the active dosing groups; Test type: Non-Inferiority or Equivalence — The non-inferiority was established if the lower limit of the one-sided, 97.5% CI in the observed difference between the proportions of subjects by study drug with Complete Cure at week 52 (itraconazole 200-mg tablets minus itraconazole 100-mg capsules) was greater than -10%. No p-value was calculated for this endpoint; Wald's CI; The statistical analysis used Wald's CI with Yates' continuity correction; Wald's CI = 0.56, 97.5% CI 1-sided [lower limit -4.3]

3. Secondary Outcome: Clinical Improvement of the Target Toenail
Description: Clinical Improvement consisted of a mycological cure and an Investigator's Global Assessment (IGA) score less than or equal to 1 at week 52.
  The Investigator's Global Assessment (IGA) assesses the overall severity of onychomycosis on the target toenail and takes into consideration, onycholysis, hyperkeratosis and percent nail involvement.
  0 = Clinical Cure: No evidence of onychomycosis.
  1 = Clinical Improvement: Minimal evidence of onychomycosis. 2 = Mild: ≤25% dystrophy and/or onycholysis. 3 = Moderate: ≤50% dystrophy with onycholysis. 4 = Severe: >50% dystrophy with onycholysis.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Groups:
- Itraconazole Capsules: Itraconazole 100mg capsules
Arm/Group | Itraconazole Tablets | Itraconazole Capsules
Number analyzed (Participants) | 593 | 590
percentage of participants | 33.7 | 29.3
Statistical Analysis 1: Comparison: Itraconazole Tablets vs Itraconazole Capsules; The test for demonstrating non-inferiority was based on a margin of 10%. Thus, non-inferiority was established if the lower limit of the one-sided, 97.5% CI in the observed difference between the proportions of subjects by study drug with Complete Cure at week 52 (itraconazole 200-mg tablets minus itraconazole 100-mg capsules) was greater than -10%. The non-inferiority analysis was restricted to the active dosing groups; Test type: Non-Inferiority or Equivalence — The assumption was that the Complete Cure rate at week 52 was 35% for the active dosing groups, a sample size of 552 ITT subjects per active group would have had a 93% power for testing the proportion of subjects with Complete Cure. These computations assumed a non inferiority margin of 10% and a one-sided significance level of 0.025. Power computations were performed using nQuery Advisor, Version 5.0; p < 0.001, Wald's CI; The statistical analysis used Wald's CI with Yates' continuity correction; Mean Difference (Final Values) = 10, 97.5% CI 1-sided [lower limit -1.1]

4. Secondary Outcome: Clinical Improvement Compared to Placebo
Description: Clinical Improvement consisted of a mycological cure and an Investigator's Global Assessment (IGA) score less than or equal to 1 at week 52.
  The Investigator's Global Assessment(IGA)assesses the overall severity of onychomycosis on the target toenail and takes into consideration, onycholysis, hyperkeratosis and percent nail involvement.
  0 = Clinical Cure: No evidence of onychomycosis.
  1 = Clinical Improvement: Minimal evidence of onychomycosis. 2 = Mild: ≤25% dystrophy and/or onycholysis. 3 = Moderate: ≤50% dystrophy with onycholysis. 4 = Severe: >50% dystrophy with onycholysis.
Time Frame: 12 months
Population: Intent to treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole Tablets | Placebo Tablets
Number analyzed (Participants) | 593 | 198
percentage of participants | 33.7 | 2
Statistical Analysis 1: Comparison: Itraconazole Tablets vs Placebo Tablets; The superiority analysis was restricted to the itraconazole 200-mg tablets and placebo tablets dosing groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; This was stratified by analysis center

ADVERSE EVENTS:
Time Frame: AEs and SAES are reported for the 12 week treatment period. SAEs are reported for both the treatment & follow-up periods in the Additional Description section.
Description: During the follow-up period, 20 subjects (10, 9, and 1 in the itraconazole 200-mg tablet, itraconazole 100-mg capsule, and placebo tablet dosing groups, respectively) reported SAEs. Because 1 subject experienced a SAE in both periods of the study, 25 individual subjects experienced SAEs during the course of the trial.
Groups:
- Itraconazole Tablets - Treatment Period: Itraconazole 200mg tablets Adverse events that occurred during the Treatment Period are reported here.
- Itraconazole Capsules: Itraconazole 100mg capsules Adverse events that occurred during the Treatment Period are reported here.
- Placebo Tablets: Adverse events that occurred during the Treatment Period are reported here.
- Itraconazole Tablets - Follow-up Period; Itraconazole Capsules - Follow-up Period; Placebo Tablets - Follow-up Period: Adverse events that occurred during the follow-up (no treatment) period are reported here.
Arm/Group | Itraconazole Tablets - Treatment Period | Itraconazole Capsules | Placebo Tablets | Itraconazole Tablets - Follow-up Period | Itraconazole Capsules - Follow-up Period | Placebo Tablets - Follow-up Period
Serious Adverse Events (participants affected / at risk) | 2/582 | 2/581 | 2/191 | 10/535 | 9/515 | 1/168
Other Adverse Events (participants affected / at risk) | 19/582 | 16/581 | 6/191 | 19/535 | 36/515 | 8/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itraconazole Tablets - Treatment Period (N=582) | Itraconazole Capsules (N=581) | Placebo Tablets (N=191) | Itraconazole Tablets - Follow-up Period (N=535) | Itraconazole Capsules - Follow-up Period (N=515) | Placebo Tablets - Follow-up Period (N=168)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carteroid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glioblatoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cenll lung caner stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itraconazole Tablets - Treatment Period (N=582) | Itraconazole Capsules (N=581) | Placebo Tablets (N=191) | Itraconazole Tablets - Follow-up Period (N=535) | Itraconazole Capsules - Follow-up Period (N=515) | Placebo Tablets - Follow-up Period (N=168)
Hypoacusis (Ear and labyrinth disorders) | 19 (19) | 16 (16) | 6 (6) | 19 (19) | 36 (36) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.